CLINICAL TRIAL: NCT05995522
Title: Effect of Vitamin K2 Supplementation and Its Association With Osteocalcin Serum Levels, Leptin, Th1/Th2 Cytokine Profile, and Cardiovascular Risk in Young Mexican Adults With Overweight and Obesity
Brief Title: Effect of Vitamin K2 Over Osteocalcin, Leptin, Cytokines, and Cardiovascular Risk in Young Adults With Overweight and Obesity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Guadalajara (Other)
Responsible Party: Principal Investigator, Andrés López Quintero, Associate Professor B, University of Guadalajara
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CI-00421
Record Dates: First submitted 2023-08-08; First posted 2023-08-16 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Overweight and Obesity; Cardiometabolic Risk Factors
Keywords: Vitamin K; Overweight and Obesity; Cardiometabolic Risk Factors
MeSH Terms: conditions — Overweight; Obesity | interventions — Vitamin K 2; Starch

STUDY DESIGN:
Intervention Model Description: Clinical trial parallel design. Two groups with intervention, one with supplementation and other with placebo
Who Masked: Participant, Investigator
Masking Description: All participants were given an identical vial, with an invention similar in shape, color, and consistency.
  The groups were named group A and group B.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Supplementation arm (Experimental): Vitamin K2
  Interventions: Dietary Supplement: Vitamin K2
- Placebo arm (Placebo Comparator): Cornstarch
  Interventions: Other: Cornstarch

INTERVENTIONS:
Dietary Supplement: Vitamin K2 — 100 µg per day for 90 days
  Other Names: Nutricost Menaquinone-4 100 µg
  Arms: Supplementation arm
Other: Cornstarch — 500 mg per day for 90 days
  Arms: Placebo arm

SUMMARY:
The goal of this clinical trial is to compare de effect of vitamin K2 in young adults with overweight or obesity. The main questions to answer are:

What is the effect of Vitamin K2 supplementation on methylation, serum concentration of ucOC, cOC, Gas6, leptin, inflammatory markers, cardiometabolic risk factors, and cardiovascular risk in overweight or obese young adults? Participants will be assigned to one of two intervention groups where they will consume Vitamin K2 100 µg per day or cornstarch 500 mg per day for 90 days.

If there is a comparison group: Investigators will compare the supplementation group (Vitamin K2) with the placebo group (cornstarch) to see if vitamin K2 supplementation modifies methylation, increases serum vitamin K, osteocalcin, growth arrest-specific 6 protein serum concentration, decreases serum leptin concentration, inflammatory markers and reduces cardiometabolic risk factors and cardiovascular risk.

DETAILED DESCRIPTION:
Study Overview To meet the objectives of the project, two groups will be compared, one that will be supplemented with vitamin K and another of patients who will receive corn starch as a placebo. Patients are going to have a follow up during 3 months with periodic evaluations every 30 days.

This is a double-blind study, it is achieved by maintaining similarities in appearance, taste and smell between the treatments that will be delivered in the same vials, with same number of pills and identical in shape, color and consistency for each study group.

Patient recruitment will take place by disseminating information through physical and social media, once potential participants have been identified, they will be contacted and informed about the project, and if they decide to participate in the study, they will be asked to sign the informed consent.

Simple randomization will be performed using R software to assign participants to one of the study groups. A clinical history, anthropometric measurements and blood sampling shall be applied.

Nutritional recommendations based on the position of the Academy of Nutrition and Dietetics for the treatment of overweight and obesity and the healthy eating plate of Harvard University will be given. An appointment is to be scheduled every 30 days in order to provide the supplementation and follow-up. At the end, the pertinent statistical analyzes will be carried out.

Notification of adverse effects will be made in each of the sessions, in addition to this the participants will have the contact of the researchers to notify any anomaly.

Sample's size calculation

The sample size was calculated using the statistical formula for the comparison of two means. This estimate was made using the following formula:

n=2(Zα+Z[1-β]2xSD2/d2

Where:

n= sample size required in each group SD= standard deviation of the effect Zα: to the value of Z for a confidence level of 95% Z[1-β}: to the value of Z for a statistical power of 80% D= effect size A total of 19.72 patients per group were obtained. Considering a 20% loss, 24 patients are needed per study group.

Ethical considerations The study was approved by the Biosafety committee, research ethics committee and research committee of the University Center for Health Sciences, University of Guadalajara: CI-00421. The committees of the University have the authority to monitor and audit the study at any of its stages once it has been approved.

Objetives General objective Evaluate the effect of vitamin K2 supplementation on methylation, the serum concentration of total vitamin K, osteocalcin, growth arrest-specific 6 protein, leptin, inflammatory markers, cardiometabolic risk factors and cardiovascular risk in young Mexican adults with overweight or obesity.

Specific objectives

1. Compare the baseline variables between groups.
2. Compare the variable changes across the time within groups
3. Compare the variable changes across the time between groups

Statistical analysis The Shapiro-Wilk normality test is performed to determine whether the analysis will require parametric or non-parametric tests. Qualitative variables will be expressed as frequencies and percentages, while quantitative variables will be expressed as mean and standard deviation in parametric data or medians and ranges in non-parametric data.

Specific objective 1 Statistical technique T-student for independent samples if it has a normal distribution or by U-Mann Whitney for independent samples if it does not have a normal distribution

Specific objective 2 Variables with two measures Statistical technique T-student for paired samples if it has a normal distribution or the Wilcoxon signed-rank test if it does not have a normal distribution

Variables with more than two measures Statistical technique Repeated measures ANOVA if it has a normal distribution or the Friedman Test if it does not have a normal distribution

Specific objective 3 Statistical technique The effect size of the groups is compared with T-student for independent samples if it has a normal distribution or by U-Mann Whitney for independent samples if it does not have a normal distribution

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index greater than 25 kg/m2 and less than 40 kg/m2
* That they agree to participate in the study voluntarily and informed and sign the informed consent

Exclusion Criteria:

* People with self-reported diagnosis of chronic kidney, gastrointestinal or systemic disease
* Use of bile acid sequestrants drugs, insulin, glucocorticoids, contraceptives, bisphosphonates, thiazides, levetiracetam, thiazolidinediones, anticoagulants or estrogenic drugs and vitamin D, vitamin K, vitamin A, vitamin E, omegas or calcium supplements
* Patients who are on a hypocaloric or low-fat diet
* Self-reported pregnancy

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2023-09-01 (Actual); Primary Completion 2023-11-30 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Osteocalcin serum concentration | Baseline and after 90 days of intervention
  ng/dL
Vitamin K serum concentration | Baseline and after 90 days of intervention
  ng/dL
Leptin serum concentration | Baseline and after 90 days of intervention
  ng/dL
Tumour Necrosis Factor alpha serum concentration | Baseline and after 90 days of intervention
  pg/mL
Interleukin-1 Beta serum concentration | Baseline and after 90 days of intervention
  pg/mL
Interleukin-6 serum concentration | Baseline and after 90 days of intervention
  pg/mL
Interleukin-4 serum concentration | Baseline and after 90 days of intervention
  pg/mL
Interleukin-10 serum concentration | Baseline and after 90 days of intervention
  pg/mL
Cardiovascular risk | Baseline, after 30, 60 and 90 days of intervention
  percentage
LEP gene methylation | Baseline and after 90 days of intervention
  Methylated or unmethylated

SECONDARY OUTCOMES:
Growth arrest-specific 6 protein serum concentration | Baseline and after 90 days of intervention
  ng/ml
Global methylation | Baseline and after 90 days of intervention
  percentage
Atherogenic indices | Baseline and after 90 days of intervention
  Value
Triglycerides serum concentration | Baseline and after 90 days of intervention
  mg/dL
Total cholesterol serum concentration | Baseline and after 90 days of intervention
  mg/dL
HDL cholesterol serum concentration | Baseline and after 90 days of intervention
  mg/dL
LDL cholesterol serum concentration | Baseline and after 90 days of intervention
  mg/dL
VLDL cholesterol serum concentration | Baseline and after 90 days of intervention
  mg/dL
Glucose serum concentration | Baseline and after 90 days of intervention
  mg/dL
Blood pressure | Baseline, after 30, 60 and 90 days of intervention
  mmHg
Insulin serum concentration | Baseline and after 90 days of intervention
  µIU/ml
Weight | Baseline, after 30, 60 and 90 days of intervention
  kg
Body mass index | Baseline, after 30, 60 and 90 days of intervention
  kg/m2
Waist circumference | Baseline, after 30, 60 and 90 days of intervention
  cm
Hip circumference | Baseline, after 30, 60 and 90 days of intervention
  cm
Fat mass | Baseline, after 30, 60 and 90 days of intervention
  kg
% fat | Baseline, after 30, 60 and 90 days of intervention
  percentage
Lean mass | Baseline, after 30, 60 and 90 days of intervention
  kg
Estimated energy consumption | Baseline, after 30, 60 and 90 days of intervention
  kcal/day
Estimated protein consumption | Baseline, after 30, 60 and 90 days of intervention
  grams/day
Estimated carbohydrates consumption | Baseline, after 30, 60 and 90 days of intervention
  grams/day
Estimated fat consumption | Baseline, after 30, 60 and 90 days of intervention
  grams/day
Estimated vitamin K consumption | Baseline, after 30, 60 and 90 days of intervention
  μg/day

CONTACTS AND LOCATIONS:
Overall Officials: Andrés López Quintero, PhD, Principal Investigator
Locations (1):
- University of Guadalajara, Guadalajara, Jalisco, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Aguayo-Ruiz JI, Garcia-Cobian TA, Pascoe-Gonzalez S, Sanchez-Enriquez S, Llamas-Covarrubias IM, Garcia-Iglesias T, Lopez-Quintero A, Llamas-Covarrubias MA, Trujillo-Quiroz J, Rivera-Leon EA. Effect of supplementation with vitamins D3 and K2 on undercarboxylated osteocalcin and insulin serum levels in patients with type 2 diabetes mellitus: a randomized, double-blind, clinical trial. Diabetol Metab Syndr. 2020 Aug 18;12:73. doi: 10.1186/s13098-020-00580-w. eCollection 2020. PMID 32831908